CLINICAL TRIAL: NCT03652805
Title: Phase 1/2a, Multi-center, Open-Label, Dose-escalating Study to Assess Safety, Tolerability, and Pharmacokinetics of Intravenously Administered IPL344 for The Treatment of Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study of IPL344 in the Treatment of ALS Patients
Acronym: ALS
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was suspended due to IPL344 shortage and may resume once drug supply is available.
Sponsor: Immunity Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101/ 2
Record Dates: First submitted 2018-08-13; First posted 2018-08-29 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPL344 (Experimental): IPL344 will be administered Intravenously on a daily basis. The dose range of IPL344 is 1.7-3.2 mg/kg
  Interventions: Drug: IPL344

INTERVENTIONS:
Drug: IPL344 — The study is designed to determine the tolerability, safety and PK of IPL344 administered I.V. once a day for 28 days and to identify the maximum tolerated dose.
  All patients enrolled will have a documented history of ALS disease prior to study enrollment.
  Treatment will start with 1.7mg/kg with dose escalation by 0.5 mg/kg every 3-4 days and will increase to the maximum dose of 3.2mg/kg. Day 1 to Day 28 patients will be on active treatment.
  After completion of 28 treatment days, participants who will choose to continue treatment (at the investigator's discretion), will be enrolled in a follow-up study. Participants that discontinue treatment after Day 28 will be followed up by a nurse phone call and return to the clinic for a final visit on Day 56 from the first dose.

SUMMARY:
This is a prospective, open-label, phase 1/2a study, dose escalation, to evaluate tolerability, safety, and PK of I.V. administered IPL344 in participants with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
The study is designed to determine the tolerability, safety and PK of IPL344 administered I.V. once a day for 28 days and to identify the maximum tolerated dose.

All patients enrolled will have a documented history of ALS disease prior to study enrollment.

Treatment will start with 1.7mg/kg with dose escalation by 0.5 mg/kg every 3-4 days and will increase to the maximum dose of 3.2mg/kg. Day 1 to Day 28 patients will be on active treatment.

After completion of 28 treatment days, participants who will choose to continue treatment (at the investigator's discretion), will be enrolled in a follow-up study. Participants that discontinue treatment after Day 28 will be followed up by a nurse phone call and return to the clinic for a final visit on Day 56 from the first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ages ≥18 to 80 years
2. Consenting participants fulfilling the El Escorial criteria for probable and definite ALS (sporadic and familial)
3. Participant has ALSFRS-R score >20, the latest ALSFRS-R test should be no more than 6 weeks before screening visit, AND:

   1. a disease progression rate greater than 0.55 ALSFRS-R point per month on average, over at least 4 months, prior to the latest ALSFRS-R test OR
   2. a decline of at least 3 points in ALSFRS-R score within the last 4 months prior to the latest ALSFRS-R test
4. Previous data of Force Vital Capacity (FVC) of ≥60% at least 3 months before screening and not more than 12 months.
5. Written informed consent consistent with ICH-GCP and local laws, signed prior to any study procedures being performed.
6. BMI 18.5 to 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg.
7. If taking riluzole or edaravone, the participant must be on a stable dose for ≥30 days prior to Day 1 and expected to remain at that dose until the final study visit.
8. Medically able to undergo the study procedures, and to adhere to the visit schedule at the time of study entry.
9. Medically is able and willing to undergo placement and maintain a central venous catheter as determined by the investigator.
10. Participant has a competent caregiver or qualified individual who can and will be responsible for the administration of study drug and reporting home activities.
11. Geographic accessibility to the study site
12. Females must not be lactating or pregnant at Screening, as documented by a negative beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG].
13. Women of child-bearing potential or males whose partners are women of child-bearing potential use an effective method of contraception throughout the trial.

Exclusion Criteria:

1. Concurrent therapy that, in the PI's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
2. Co-existing psychiatric disorder excluding a depression disorder occurred after ALS diagnosis.
3. Participant is a respiratory dependent.
4. Subjects with a significant pulmonary disorder not attributed to ALS.
5. Slow Vital Capacity (SVC) <60.
6. Presence of any other condition or circumstance that, in the judgment of the Investigator, might contraindicate or increase the risk to the participant or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
7. History of HIV, positive HBV or HCV serology.
8. Participants suffering from significant cardiac, or any other disease that may endanger the participant or interfere with the ability to interpret the results.
9. A participant with active infections.
10. Documented active cancer.
11. Treatment with another investigational drug, biological agent, or device within 2 months of the first dose, or investigational cell therapy within 6 months of the first dose.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) and serious adverse events (SAEs) Reporting | (up-to Day 56)
  All AEs will be recorded, whether considered minor or serious, drug-related or not
Maximum Tolerated Dose (MTD) | Study treatment duration (Day 1 -28 days)
  Dose defined as the highest dose with no Dose Limiting Toxicity (DLT). DLT will be defined as a Grade ≥ 3 toxicity per participant according to Common Terminology Criteria for Adverse Events (CTCAE v5.0).

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile - Maximum Plasma Concentration (Cmax) | Pre-Dose and 5, 10, 20, 30, 45, 60 and 120 minutes after dosing
  Blood will be collected for PK testing on Day 1 prior to and after first dose and on each dose-escalation administration day and on Day 28
Pharmacokinetic (PK) profile - Area Under the Curve (AUC) | Pre-Dose and 5, 10, 20, 30, 45, 60 and 120 minutes after dosing
  Blood will be collected for PK testing on Day 1 prior to and after first dose and on each dose-escalation administration day and on Day 28
Pharmacokinetic (PK) profile - time to reach maximum plasma concentration (Tmax) | Pre-Dose and 5, 10, 20, 30, 45, 60 and 120 minutes after dosing
  Blood will be collected for PK testing on Day 1 prior to and after first dose and on each dose-escalation administration day and on Day 28
Pharmacokinetic (PK) profile - apparent terminal exponential half-life (T1/2) | Pre-Dose and 5, 10, 20, 30, 45, 60 and 120 minutes after dosing
  Blood will be collected for PK testing on Day 1 prior to and after first dose and on each dose-escalation administration day and on Day 28

OTHER OUTCOMES:
Exploratory: Biomarker testing | up-to Day 56
  Blood samples for exploratory Biomarkers (Biobanking)
Exploratory: Anti-Drug Antibody (ADA) testing | up-to Day 56
  Blood samples for Anti-Drug Antibody (Biobanking)
Exploratory: identify a marker based on the mechanism of action (MOA) | up-to Day 56
  Blood samples for future PD (Biobanking)
Changes from baseline in ALS disease progression | up-to day 56
  ALS functional rating scale-Revised (ALSFRS-R) - Questionnaire
Changes from baseline in Pulmonary Function | up-to day 56
  Measured by Vital Capacity (VC)
Changes from baseline in Muscle strength | up-to day 56
  Assessed by using a quantitative strength testing tool, Hand Held Dynamometry (HHD)
Changes from baseline in Anti-Depression effect | up-to day 56
  Evaluated by ALS Depression Inventory (ADI-12) - questionnaire
Changes from baseline in Anti-Depression effect | up-to day 56
  the Hospital Anxiety and Depression Scale (HADS) - questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center -Motor Neuron Disease Clinic, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No